CLINICAL TRIAL: NCT06394258
Title: POSE (POs Surgery Endometrial Cancer) - Phase I/II Study to Access SBRT as a Replacement for Brachytherapy in Intermediate and High Risk in Endometrial Cancer
Brief Title: POSE - POs Surgery Endometrial Cancer
Acronym: POSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Inês Antunes, Principal Investigator, Fundacao Champalimaud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POSE2
Record Dates: First submitted 2024-01-10; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Endometrial Cancer adjuvant treatment: Exclusive fractionated radiosurgery 21 Gy/3 fractions (BED10 35,7 Gy) prescribed to 100% isodose at 5 mm from the mucosa surface and 150% isodose to the mucosa surface (BED10 64,675 Gy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT to the vaginal cuff (Experimental): SBRT to the vaginal cuff
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — Stereotactic body radiotherapy to the vaginal cuff with the aim to reproduce adjuvant high dose rate (HDR) brachytherapy dose distribution by means of external beam radiotherapy in patients operated for intermediate risk endometrial carcinoma
  Other Names: Stereotactic ablative body radiotherapy (SABR)

SUMMARY:
This phase I/II feasibility study of hypo-fractionated, image-guided Volumetric Modulated Arc Therapy (VMAT) Stereotactic Body Radiotherapy (SBRT) to the vaginal cuff in intermedium and high risk endometrial cancer. The primary endpoints are SBRT feasibility and dosimetrical reproducibility to HDR brachytherapy, inter/intra-fractional target motion assessment and toxicity rates. Secondary endpoints are quality of life measures, local control, disease free survival and overall survival.

DETAILED DESCRIPTION:
This phase I/II feasibility study of hypo-fractionated, image-guided Volumetric Modulated Arc Therapy (VMAT) Stereotactic Body Radiotherapy (SBRT) to the vaginal cuff aims to reproduce adjuvant High Dose Rate (HDR) brachytherapy dose distributions in patients operated for intermediate and high risk endometrial carcinoma. The study will employ devices to accurately reproduce pelvic anatomy and mitigate target motion and will make use of real-time on-line tracking. Eligible patients will receive three SBRT sessions to a prescription dose of 7 Gy to the vaginal cuff (with 4 to 7 days interval). SBRT will start within 4 to 8 weeks post-hysterectomy. The study will enroll a total of 30 patients. After treatment, patients will be followed-up at 3 months (+/- 6 weeks), at 6 (+/- 6 weeks) and every 6 months (+/- 6 weeks) thereafter for a total of 2 years. The duration of accrual in the study will be up to 3 years. Toxicity and outcome will be compared to published data on the standard modality of care (HDR brachytherapy). Patients' quality of life measures will be collected with validated questionnaires at the baseline and during follow up. Recurrence rates and survival data will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Pathology proven adenocarcinoma of the endometrium
* National Comprehensive Cancer Network (NCCN) intermediate and high risk
* Unstaged patients with < 50% myometrium invasion;
* Age ≥ 18;
* World health organization - Eastern Cooperative Oncology Group (WHO-ECOG) performance status 0-2 or Karnofsky performance status (KPS) ≥ 70;
* Hemoglobin ≥ 8.0 g/dl; white blood cells count (WBC) ≥ 1,500/mm3 ; Platelets ≥ 40,000 cells/mm3 .
* Signed informed consent

Exclusion Criteria:

* Evidence of post-surgical macroscopic residual disease;
* Patients with anatomical incompatibility with online tracking device;
* Psychiatric conditions;
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years;
* Prior radiation therapy to the pelvis that would result in overlap of radiation therapy fields;
* Severe active co-morbidities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Dosimetric Feasibility of vaginal cuff SBRT | through study completion, an average of 3 year
  Fulfillment of protocol dosimetrical endpoints and constraints; physician assessment of complications (CTCAE V3.0) at specific time points during follow up (2 weeks, 3 and 6 months, then every 6 months until the end of the 3rd year, then annually until the end of the 5th year)
Reproducibility of vaginal cuff SBRT | Accuracy of treatment delivery will be measured during the 15 minutes of treatment delivery time
  Anatomical accuracy will be confirmed with image guided (CBCT) and online tracking will guarantee a limit of 2mm threshold
Inter/intra fractional target motion | during the 15 minutes of treatment delivery time
  3D deviations recorded in CBCT images and electromagnetic recording
Adverse Events | through study completion, an average of 5 years
  Treatment related side effects based on CTCAE V3.0

SECONDARY OUTCOMES:
Quality of life metrics | through study completion, an average of 5 years
  change from baseline in European Organisation for Research and Treatment of Cancer quality of life questionnaire C30
Quality of life metrics | through study completion, an average of 5 years
  change from baseline in European Organisation for Research and Treatment of Cancer quality of life questionnaire quality of life questionnaire N24
Quality of life metrics | through study completion, an average of 5 years
  scoring more than 12 points in Hospital Anxiety and Depression Scale (HADS)
Local control | through study completion, an average of 5 years
  Free from loco-regional relapse
Distant Relapse | through study completion, an average of 5 years
  Free from distant relapse

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Greco, Study Director — Radiotherapy Director Unit
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No